CLINICAL TRIAL: NCT06860022
Title: Sentence Shaping: Written Language Intervention for Deaf and Hard of Hearing Middle Schoolers
Brief Title: Sentence Shaping - DHH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Adriana M. Valtierra, Principal Investigator, Vanderbilt University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 240927
Record Dates: First submitted 2025-02-27; First posted 2025-03-05 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-10

CONDITIONS: Hearing Loss, Bilateral
MeSH Terms: conditions — Hearing Loss, Bilateral

STUDY DESIGN:
Intervention Model Description: Single-case multiple probe across participants
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Shape coding (Experimental): Intervention will be introducing and utilizing Shape Coding to construct sentences.
  Interventions: Behavioral: Shape Coding

INTERVENTIONS:
Behavioral: Shape Coding — Intervention will include introducing and reviewing the relevant shapes from Shape Coding and the order in which the shapes go in a sentence. The researcher will then model how to put the word tiles in order according to the shapes. Next the researcher and student work together to construct sentences. The student is then given the opportunity to independently construct sentences using the word tiles and Shape Coding. At the end of instruction, the researcher and student review the shapes and the student has the opportunity to independently construct sentences without shape coding.

SUMMARY:
The proposed research addresses a long-standing and important challenge of improving literacy skills of children who are deaf and hard of hearing, a historically under researched group. The investigators aim to leverage shape coding - an empirically validated intervention approach for constructing sentences in spoken English - for improving how efficiently children who are deaf and hard of hearing learn to correctly construct sentences in written English. To advance the promising yet underutilized research on shape coding, the investigators complete the next logical step of applying the visual supports provided with shape coding to written language for deaf and hard of hearing children. Shape coding has been effective for teaching sentence structure in spoken English to children with language disabilities and has recently been applied to sentence structure in American Sign Language with deaf and hard of hearing children. Intervention involving shape coding is predicted to result in increased accuracy of word order in sentences in written English because deaf and hard of hearing children often benefit from visual information. The investigators will accomplish this aim using single case multiple probe across participants design studies with 30 fifth through eighth grade children who are deaf and hard of hearing. The knowledge gained will guide language and literacy intervention for children who are deaf and hard of hearing.

ELIGIBILITY:
Inclusion Criteria:

* Children in grades five through eight
* deaf or hard of hearing
* use spoken English and American Sign Language (ASL)
* bilateral hearing loss
* the ability to read and understand the grammatical structures of interest
* already be writing sentences, but demonstrate errors in word order and/or grammar.

Exclusion Criteria:

* diagnosis of dyslexia
* uncorrected vision impairment (i.e., identified vision loss without use of corrective lenses that interferes with eligibility evaluation tasks)
* evidence of severe motor impairment (i.e., insufficient motor skills to complete eligibility evaluation tasks independently).

Ages: 9 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2025-08-28 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Proportion of children for whom the intervention is successful | Baseline to up to 8 weeks maximum
  The investigators will calculate the proportion of children for whom the intervention is successful, defined as at least 80% accuracy for 3 consecutive data collection days.

SECONDARY OUTCOMES:
Proportion of children that generalize targeted skill to unpracticed words within targeted structure | Baseline to up to 8 weeks maximum
  The investigators will calculate the proportion of children that generalize the targeted skill to novel/unpracticed words within the targeted structure.
Proportion of children that generalize targeted skill to unpracticed modality within targeted structure | Baseline to up to 8 weeks maximum.
  The investigators will calculate the proportion of children that generalize the targeted skill to an unpracticed modality (i.e., writing, typing) using practiced words within the targeted structure.
Proportion of children that maintain targeted skill after intervention has ended | Begins no more than 2 weeks after intervention phase ends; lasts up to 3 weeks
  The investigators will calculate the proportion of children that maintain higher percent accuracy after intervention is removed compared to baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Undecided